CLINICAL TRIAL: NCT01231581
Title: A Randomized, Double-Blind Placebo-Controlled Phase II Study of the MEK Inhibitor GSK1120212 Plus Gemcitabine vs Placebo Plus Gemcitabine in Subjects With Metastatic Pancreatic Cancer
Brief Title: Study of GSK1120212 Plus Gemcitabine vs Placebo Plus Gemcitabine in Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113487
Record Dates: First submitted 2010-08-30; First posted 2010-11-01 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — trametinib; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GSK1120212 plus Gemcitabine (Experimental): GSK1120212 administered orally plus gemcitabine IV
  Interventions: Drug: GSK1120212; Drug: Gemcitabine
- Placebo plus Gemcitabine (Active Comparator): Placebo administered orally plus gemcitabine IV
  Interventions: Drug: Gemcitabine; Drug: Placebo

INTERVENTIONS:
Drug: GSK1120212 — administered orally starting on day 1 followed by a continuous daily dosing of 2.0 mg
  Arms: GSK1120212 plus Gemcitabine
Drug: Gemcitabine — Intravenous gemcitabine infused over 30 minutes weekly for 7 weeks followed by one week of rest from treatment. Subsequent cycles will consist of 1000 mg/m2 intravenous infusion over 30 minutes on days 1, 8, and 15 followed by 1 week of rest from treatment for each 28-day treatment period.
Drug: Placebo — administered orally starting on day 1 followed by a continuous daily dosing of 2.0 mg
  Arms: Placebo plus Gemcitabine

SUMMARY:
GSK1120212 is a potent and highly selective inhibitor of MEK phosphorylation and kinase activity and has demonstrated potent anti-proliferative activity against human pancreatic cancer cell lines. This study is a Phase II, randomized placebo-controlled trial of the MEK inhibitor GSK1120212 plus gemcitabine vs. placebo plus gemcitabine in subjects with metastatic pancreatic cancer. Eligible subjects will receive intravenous gemcitabine with oral GSK1120212 or placebo. Therapy will continue until treatment discontinuation criteria are met. The primary objective will be to compare the overall survival of subjects in the GSK1120212 plus gemcitabine arm vs. subjects in the placebo plus gemcitabine arm. Secondary objectives include comparison of progression free survival, overall response rate, and duration of response between the two arms. Exploratory research objectives include the evaluation of population pharmacokinetics as well as blood and tissue based biomarkers. Safety will also be monitored throughout dosing.

Once the determined number of survival events has occurred, if subjects are eligible, they will have the option to enter MEK114375, an open-label, Phase Ib rollover study of GSK1120212 monotherapy or GSK1120212 in combination with other anti-cancer treatments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Histologically or cytologically confirmed diagnosis of metastatic (Stage IV) adenocarcinoma of the pancreas with measurable or non-measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Performance status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale
* All prior treatment related toxicities must be Common Terminology Criteria for Adverse Events (CTCAE) (Version 4.0) ≤ Grade 1 (except alopecia) at the time of randomization
* Adequate baseline organ function
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels

Exclusion Criteria:

* Prior systemic therapy (i.e., chemotherapy, immunotherapy, hormone therapy, , targeted therapy or any investigational anti-cancer drug) for metastatic pancreatic adenocarcinoma.

(Prior treatment with 5-FU based or gemcitabine administered as a radiation sensitizer during and up to 4 weeks after radiation therapy is allowed. Prior systemic chemotherapy in the adjuvant setting is allowed ; however, prior therapy with gemcitabine is allowed only if tumor recurrence occurred at least 6 months after completing the last dose of gemcitabine)

* History of another malignancy. Exception: Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible. Subjects with second malignancies that are indolent or definitively treated may be enrolled. Consult GSK Medical Monitor if unsure whether second malignancies meet requirements specified above
* Any serious and/or unstable pre-existing medical (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator or GSK Medical Monitor
* History of interstitial lung disease or pneumonitis
* History or current evidence / risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR)
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression
* History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Seoul, South Korea
- Taiwan (3):
  - GSK Investigational Site, Gueishan Township,Taoyuan County
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei

REFERENCES:
- [Derived] Infante JR, Somer BG, Park JO, Li CP, Scheulen ME, Kasubhai SM, Oh DY, Liu Y, Redhu S, Steplewski K, Le N. A randomised, double-blind, placebo-controlled trial of trametinib, an oral MEK inhibitor, in combination with gemcitabine for patients with untreated metastatic adenocarcinoma of the pancreas. Eur J Cancer. 2014 Aug;50(12):2072-81. doi: 10.1016/j.ejca.2014.04.024. Epub 2014 Jun 7. PMID 24915778

RESULTS

PARTICIPANT FLOW:
Groups:
- Trametinib + Gemcitabine: Participants received 2 milligrams (mg) trametinib orally once daily in combination with 1000 mg/m^2 of gemcitabine given as intravenous (IV) infusion over 30 minutes (min). In the first cycle, gemcitabine was infused weekly for 7 weeks followed by a week of rest from treatment and then subsequent cycles on Day 1, 8, and 15 followed by 1 week of rest from treatment for each 28-day treatment cycle until progressive disease (PD), unacceptable toxicity, or permanent discontinuation from study treatment for any reason.
- Placebo + Gemcitabine: Participants received placebo orally once daily in combination with 1000 mg/m^2 of gemcitabine given as IV infusion over 30 min. In the first cycle, gemcitabine was infused weekly for 7 weeks followed by a week of rest from treatment and then subsequent cycles on Day 1, 8, and 15 followed by 1 week of rest from treatment for each 28-day treatment cycle until PD, unacceptable toxicity, or permanent discontinuation from study treatment for any reason.
Period: Overall Study
Arm/Group | Trametinib + Gemcitabine | Placebo + Gemcitabine
Started | 80 | 80
Ongoing | 1 (Participant is continuing treatment with trametinib and gemcitabine under roll over study MEK114375.) | 0
Completed | 0 | 0
Not Completed | 80 | 80
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Study Closed/Terminated | 6 | 5
Not completed — Death | 65 | 64
Not completed — Ongoing | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trametinib + Gemcitabine | Placebo + Gemcitabine | Total
Number analyzed (Participants) | 80 | 80 | 160
Age Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (10.35) | 62.2 (9.56) | 62.3 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 34 | 75
  Male | 39 | 46 | 85
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 50 | 59 | 109
  Asian - East Asian Heritage | 24 | 13 | 37
  African American Africa | 6 | 5 | 11
  Asian - Central/South Asian Heritage | 0 | 1 | 1
  Asian - South East Asian Heritage | 0 | 1 | 1
  White - Arabic/North African Heritage | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization until death due to any cause. For the analysis of overall survival, the last date of known contact was used for those participants who were not dead at the time of analysis; such participants were considered censored.
Time Frame: From randomization until death due to any cause or until the data cutoff of 15-March-2013 (up to 24 months)
Population: Intent-to-Treat (ITT) Population: all randomized participants regardless of whether or not treatment was administered
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trametinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 80 | 80
months | 8.4 [7.8 to 10.3] | 6.7 [5.3 to 9.9]
Statistical Analysis 1: Comparison: Trametinib + Gemcitabine; Test type: Superiority or Other; p = 0.352, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.66 to 1.32] — Hazard ratios are estimated using a Pike estimator

2. Secondary Outcome: Progression-free Survival (PFS) as Assessed by the Investigator
Description: PFS is defined as the time from randomization until the earliest date of radiological PD or death due to any cause. PD was based on radiographic or photographic evidence, and assessments were made by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 millimeters (mm). PD was also based on unequivocal progression of existing non-target lesions. If the participant received subsequent anti-cancer therapy prior to the date of documented progression or death, or did not have a documented date of progression or death, PFS was censored at the last adequate assessment.
Time Frame: From randomization until disease progression (PD) or death due to any cause or until the data cutoff of 17-April-2012 (up to 15 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Trametinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 80 | 80
weeks | 16.1 [14.0 to 23.4] | 15.1 [8.6 to 21.7]

3. Secondary Outcome: Number of Participants With an Investigator-assessed Best Response, With or Without Confirmation, of Complete Response (CR) or Partial Response (PR)
Description: CR is defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes must be <10 mm in the short axis. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g., percent change from baseline). CR and PR were evaluated by the Investigator using standard criteria (RECIST version 1.1). Confirmation of response was not required.
Time Frame: From randomization until disease progression or death due to any cause or until the data cutoff of 17-April-2012 (up to 15 months)
Population: Measurable Disease (MD) Population: all randomized participants regardless of whether or not treatment was administered who had measurable disease at baseline
Measure: Number; unit: participants
Arm/Group | Trametinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 77 | 77
participants
  CR | 1 | 0
  PR | 16 | 14

4. Secondary Outcome: Investigator-Assessed Duration of Response
Description: Duration of response is defined, for the subset of participants with a CR or PR, as the time from the first documented evidence of CR or PR until the first documented disease progression or death due to any cause. CR is defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes must be <10 mm in the short axis. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g., percent change from baseline). PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start).
Time Frame: From the first documented CR or PR until disease progression or death due to any cause or until the data cutoff of 17-April-2012 (up to 13 months)
Population: MD Population. Duration of response was assessed for only those participants with a CR or PR.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Trametinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 17 | 14
Weeks | 23.9 [9.0 to 28.9] | 16.1 [8.3 to NA] — There were too few events to provide an estimable upper limit of the confidence interval.

5. Secondary Outcome: Number of Participants With Any Adverse Event (AE) and Any Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury. Per protocol other events were considered SAEs like symptomatic left ventricular ejection fraction (LVEF) decreases or cases of central serous retinopathy (CSR) or retinal vein occlusion (RVO). AE and SAE data were collected from the start of the first dose of study treatment and continued until 28 days following discontinuation of the study treatment or death. Refer to the general AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From the start of the first dose of study treatment until 28 days following discontinuation of the study treatment or until the data cutoff of 15-March-2013 (up to 21 months)
Population: Safety Population: all participants who were randomized and took at least one dose of study medication. This population was based on the actual treatment received, if it differed from that to which the participant was randomized.
Measure: Number; unit: participants
Arm/Group | Trametinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 80 | 80
participants
  Any AE | 80 | 80
  SAE | 42 | 37

6. Secondary Outcome: Number of Participants (Par.) With a Worst-case Change to Grade 3 or Grade 4 From Baseline Grade in Chemistry Parameters
Description: A grading (severity) scale is provided for each laboratory toxicity. Grade refers to the severity of the toxicity. The Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 displays Grades 1 through 5 based on the general guideline: Grade 1, mild toxicity; Grade 2, moderate toxicity; Grade 3, severe toxicity; Grade 4, life-threatening or disabling toxicity; Grade 5, death related to toxicity.
Time Frame: From the start of the first dose of study treatment until 28 days following discontinuation of the study treatment or until the data cutoff of 17-April-2012 (up to 17 months)
Population: Safety Population. Only those par. with laboratory values for worst-case on therapy were analyzed. The same par. were not necessarily analyzed for each laboratory parameter; thus, the number of par. analyzed reflects all par. in the Safety Population. The number of par. analyzed for a particular parameter is included in the parameter title.
Measure: Number; unit: participants
Arm/Group | Trametinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 80 | 80
participants
  Albumin, Grade 3, n=73, 73 | 7 | 4
  Albumin, Grade 4, n=73, 73 | 0 | 0
  Alkaline Phosphatase, Grade 3, n=74, 73 | 7 | 4
  Alkaline Phosphatase, Grade 4, n=74, 73 | 0 | 0
  Alanine Amino Transferase, Grade 3, n=74, 73 | 7 | 7
  Alanine Amino Transferase, Grade 4, n=74, 73 | 0 | 0
  Aspartate Aminotransferase, Grade 3, n=73, 72 | 6 | 7
  Aspartate Aminotransferase, Grade 4, n=73, 72 | 0 | 0
  Total Bilirubin, Grade 3, n=74, 73 | 1 | 7
  Total Bilirubin, Grade 4, n=74, 73 | 0 | 1
  Calcium (hypercalcemia), Grade 3, n=73, 73 | 1 | 1
  Calcium (hypercalcemia), Grade 4, n=73, 73 | 0 | 0
  Calcium (hypocalcemia), Grade 3, n=73, 73 | 1 | 2
  Calcium (hypocalcemia), Grade 4, n=73, 73 | 0 | 0
  Creatinine, Grade 3, n=74, 75 | 0 | 0
  Creatinine, Grade 4, n=74, 75 | 1 | 0
  Glucose (hyperglycemia), Grade 3, n=74, 72 | 9 | 10
  Glucose (hyperglycemia), Grade 4, n=74, 72 | 0 | 1
  Glucose (hypoglycemia), Grade 3, n=74, 72 | 0 | 0
  Glucose (hypoglycemia), Grade 4, n=74, 72 | 1 | 0
  Potassium (hyperkalemia), Grade 3, n=74, 72 | 2 | 1
  Potassium (hyperkalemia), Grade 4, n=74, 72 | 0 | 0
  Potassium (hypokalemia), Grade 3, n=74, 72 | 4 | 1
  Potassium (hypokalemia), Grade 4, n=74, 72 | 0 | 0
  Sodium (hyponatremia), Grade 3, n=74, 74 | 5 | 3
  Sodium (hyponatremia), Grade 4, n=74, 74 | 2 | 0

7. Secondary Outcome: Number of Participants With Change From Baseline Increase to Grade 3/Grade 4 in Lab Hematology Test Measurements
Description: A grading (severity) scale is provided for each laboratory toxicity. Grade refers to the severity of the toxicity. The CTCAE version 3.0 displays Grades 1 through 5, with unique clinical descriptions of the severity for each toxicity based on the general guideline: Grade 1, mild toxicity; Grade 2, moderate toxicity; Grade 3, severe toxicity; Grade 4, life-threatening or disabling toxicity; Grade 5, death related to toxicity.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Trametinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 80 | 80
participants
  Hemoglobin (Increased), Grade 3, n=80, 79 | 3 | 0
  Hemoglobin (Increased), Grade 4, n=80, 79 | 0 | 0
  Hemoglobin (Anemia), Grade 3, n=80, 79 | 24 | 13
  Hemoglobin (Anemia), Grade 4, n=80, 79 | 0 | 0
  Lymphocytes (Increased), Grade 3, n=80, 79 | 1 | 0
  Lymphocytes (Increased), Grade 4, n=80, 79 | 0 | 0
  Lymphocytes (Decreased), Grade 3, n=80, 79 | 9 | 12
  Lymphocytes (Decreased), Grade 4, n=80, 79 | 3 | 6
  Absolute Neutrophil Count, Grade 3, n=80, 79 | 23 | 20
  Absolute Neutrophil Count, Grade 4, n=80, 79 | 7 | 10
  Platelet count, Grade 3, n=80, 79 | 11 | 10
  Platelet count, Grade 4, n=80, 79 | 1 | 4
  White Blood Cell count, Grade 3, n=80, 79 | 15 | 14
  White Blood Cell count, Grade 4, n=80, 79 | 1 | 4

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the time the first dose of study treatment was administered until 28 days following discontinuation of study treatment or until the data cutoff of 15-March-2013 (up to 21 months).
Description: SAEs and non-serious AEs were collected in the Safety Population, comprised of all participants who were randomized and took at least one dose of study medication. This population was based on the actual treatment received, if it differed from that to which the participant was randomized.
Arm/Group | Trametinib + Gemcitabine | Placebo + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 42/80 | 37/80
Other Adverse Events (participants affected / at risk) | 80/80 | 80/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trametinib + Gemcitabine (N=80) | Placebo + Gemcitabine (N=80)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 2
Sepsis (Infections and infestations) | 3 | 2
Biliary tract infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 3
Abdominal sepsis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Postoperative abscess (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 2
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 2
Jaundice (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Pyrexia (General disorders) | 8 | 2
Asthenia (General disorders) | 1 | 1
Device occlusion (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Stent malfunction (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 3
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trametinib + Gemcitabine (N=80) | Placebo + Gemcitabine (N=80)
Nausea (Gastrointestinal disorders) | 43 | 41
Vomiting (Gastrointestinal disorders) | 38 | 36
Diarrhoea (Gastrointestinal disorders) | 43 | 22
Constipation (Gastrointestinal disorders) | 23 | 20
Stomatitis (Gastrointestinal disorders) | 29 | 6
Abdominal pain (Gastrointestinal disorders) | 15 | 14
Abdominal pain upper (Gastrointestinal disorders) | 9 | 9
Abdominal distension (Gastrointestinal disorders) | 7 | 8
Ascites (Gastrointestinal disorders) | 6 | 8
Dyspepsia (Gastrointestinal disorders) | 8 | 4
Flatulence (Gastrointestinal disorders) | 3 | 7
Dry mouth (Gastrointestinal disorders) | 4 | 5
Gingival bleeding (Gastrointestinal disorders) | 4 | 0
Haemorrhoids (Gastrointestinal disorders) | 4 | 0
Fatigue (General disorders) | 30 | 30
Oedema peripheral (General disorders) | 30 | 25
Pyrexia (General disorders) | 27 | 26
Asthenia (General disorders) | 9 | 13
Chills (General disorders) | 8 | 9
Mucosal inflammation (General disorders) | 9 | 4
Influenza like illness (General disorders) | 1 | 7
Pain (General disorders) | 4 | 3
Anaemia (Blood and lymphatic system disorders) | 37 | 34
Thrombocytopenia (Blood and lymphatic system disorders) | 32 | 22
Neutropenia (Blood and lymphatic system disorders) | 28 | 22
Leukopenia (Blood and lymphatic system disorders) | 9 | 8
Lymphopenia (Blood and lymphatic system disorders) | 1 | 5
Rash (Skin and subcutaneous tissue disorders) | 38 | 20
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 10
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 12 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4
Acne (Skin and subcutaneous tissue disorders) | 6 | 1
Platelet count decreased (Investigations) | 22 | 16
Alanine aminotransferase increased (Investigations) | 12 | 16
Aspartate aminotransferase increased (Investigations) | 11 | 12
Neutrophil count decreased (Investigations) | 9 | 14
Weight decreased (Investigations) | 9 | 9
Haemoglobin decreased (Investigations) | 5 | 7
Blood alkaline phosphatase increased (Investigations) | 3 | 11
Ejection fraction decreased (Investigations) | 7 | 2
White blood cell count decreased (Investigations) | 0 | 8
Blood creatinine increased (Investigations) | 5 | 0
Blood bilirubin increased (Investigations) | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 25 | 25
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 | 4
Dehydration (Metabolism and nutrition disorders) | 5 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dizziness (Nervous system disorders) | 12 | 11
Headache (Nervous system disorders) | 6 | 10
Dysgeusia (Nervous system disorders) | 7 | 7
Tremor (Nervous system disorders) | 2 | 6
Depression (Psychiatric disorders) | 5 | 9
Insomnia (Psychiatric disorders) | 8 | 3
Anxiety (Psychiatric disorders) | 4 | 5
Deep vein thrombosis (Vascular disorders) | 6 | 4
Hypotension (Vascular disorders) | 4 | 6
Hypertension (Vascular disorders) | 2 | 6
Urinary tract infection (Infections and infestations) | 2 | 7
Paronychia (Infections and infestations) | 9 | 0
Nasopharyngitis (Infections and infestations) | 4 | 3
Cellulitis (Infections and infestations) | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4
Vision blurred (Eye disorders) | 7 | 10
Periorbital oedema (Eye disorders) | 4 | 0
Dysuria (Renal and urinary disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.